CLINICAL TRIAL: NCT05910177
Title: A Single Arm, Exploratory Clinical Study on the Neoadjuvant Treatment of Neuroendocrine Cervix Carcinoma With Camrelizumab Combined With Etoposide and Cisplatin
Brief Title: Neoadjuvant Treatment of Neuroendocrine Cervix Carcinomar With Camrelizumab Combined With Etoposide and Cisplatin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hhaixin
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma; Cervix Carcinoma
MeSH Terms: conditions — Carcinoma; Uterine Cervical Neoplasms | interventions — Etoposide; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Karelizumab combined with etoposide and cisplatin group (Experimental): The cycle dose should be strictly controlled according to the experimental design. The order of administration is as follows: Karelizumab → Cisplatin → Etoposide (with an interval of at least 30 minutes)
  Interventions: Drug: Karelizumab combined with etoposide and cisplatin

INTERVENTIONS:
Drug: Karelizumab combined with etoposide and cisplatin — Karelizumab：200 mg，ivgtt，D1，q3w； Cisplatin：75 mg/m2，ivgtt，D1，q3w； Etoposide：100 mg/m2，ivgtt，D1~3，q3w
  Other Names: Karelizumab

SUMMARY:
This study is a single arm, exploratory clinical study aimed at evaluating the efficacy and safety of karelizumab combined with etoposide and cisplatin in the neoadjuvant treatment of neuroendocrine cervix carcinoma.

DETAILED DESCRIPTION:
This study is a single arm, exploratory clinical study aimed at evaluating the efficacy and safety of karelizumab combined with etoposide and cisplatin in the neoadjuvant treatment of neuroendocrine cervix carcinoma.Following this, patients achieving complete or partial response will proceed to radical surgery and adjuvant therapy, while those with stable or progressive disease, or considered unsuitable for surgery by gynecological oncologists, will transfer to concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years ≤ Age ≤ 75 years, female patient. 2. Patients with cervical neuroendocrine carcinoma confirmed by histopathology or cytology (if mixed type carcinoma, the composition of neuroendocrine carcinoma is>60%), whose FIGO stage is stage I-II, and who can be operated according to the gynecological examination of an experienced Chief physician.

3. According to the RECIST 1.1 standard, patients have at least one measurable diameter target lesion (tumor lesion CT scan length ≥ 10mm, lymph node lesion CT scan short diameter ≥ 15mm, scan layer thickness 5mm).

4. ECOG PS 0-1 points. 5. The estimated postoperative survival time is greater than 3 months. 6. The main organs function normally and meet the following standards:

1. The blood routine test must meet the following criteria: (no blood transfusion within 14 days)

   1. HB ≥ 100g/L
   2. WBC ≥ 3 × 109/L
   3. ANC ≥ 1.5 × 109/L
   4. PLT ≥ 100 × 109/L
2. Biochemical examination must meet the following standards:

   1. BIL<1.5 times upper limit of normal value (ULN)
   2. ALT and AST<2.5ULN, GPT ≤ 1.5 × ULN
   3. Serum Cr ≤ 1ULN, endogenous creatinine clearance rate>60ml/min (Cockcroft Goult formula).

      7. Not participating in other clinical studies before and during treatment.

      8. Women of childbearing age must undergo a serum pregnancy study within 7 days before the first medication use, and the results should be negative. Female participants of childbearing age and male participants with partners of childbearing age must agree to contraception within 24 weeks after signing the informed consent form and the last administration of the study medication.

      9. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

      Exclusion Criteria:
      1. Those who have a history of chemotherapy, radiation therapy, targeted drug therapy, or immunotherapy in the past.
      2. Patients who have Contraindication to surgical treatment and chemotherapy or whose physical condition and organ function do not allow large abdominal surgery.
      3. Distant metastasis.
      4. Have any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, Uveitis, enteritis, hepatitis, hypophysitis, Vasculitis, Myocarditis, nephritis, Hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Except for Vitiligo or recovered childhood asthma/allergy patients who do not need any intervention after adulthood; Autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with a stable dose of insulin.
      5. Have a history of immune deficiency, including positive Diagnosis of HIV/AIDS, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation.
      6. Accompanied by severe heart, lung, liver, and kidney diseases; Having neurological or mental illness; Individuals with jaundice or gastrointestinal obstruction and severe infections.
      7. Pregnant or lactating women.
      8. Suffering from coronary heart disease of grade I or above, arrhythmia (including prolonged QTc interval, female>470 ms), and cardiac dysfunction.
      9. Patients with abnormal coagulation function (INR>1.5, APTT>1.5 ULN).
      10. The subject has clinical cardiovascular symptoms or diseases that cannot be well controlled, including but not limited to: (1) NYHA grade II or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias that are still poorly controlled without or after clinical intervention.
      11. Have a history of Interstitial lung disease (excluding radiation pneumonia without hormone treatment) and non infectious pneumonia.
      12. People who have been allergic to any component of Camrelizumab or any component of the study medication in the past.
      13. Researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6-month
  The proportion of participants achieving Complete Response (CR), Partial Response (PR) or Stable Disease (SD) according to RECIST1.1.

SECONDARY OUTCOMES:
Progression-free survival | 6-month
  The period between the onset of treatment and the observation of disease progression or the occurrence of death for any reason.
Disease-free survival period | 6-month
  After radical treatment (complete surgical removal of the tumor), there is no time for the disease to recur.
1 year and 3 year overall survival rates | 1 year and 3 year
  The proportion of patients who have survived for one and three years after comprehensive treatment.
1-year and 3-year progression free survival rates | 1 year and 3 year
  The probability that the patient's disease will not continue to worsen within one and three years.
1-year and 3-year disease control rates | 1 year and 3 year
  The proportion of patients with reduced or stable tumors within 1 and 3 years.
Incidence rate of adverse events | 5 years
  The ratio of the number of cases with adverse events to the total number of cases available for evaluation.
Disease control rate | 6-month
  The proportion of participants achieving Complete Response (CR), Partial Response (PR) or Stable Disease (SD) according to RECIST1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China